CLINICAL TRIAL: NCT03048123
Title: The Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy Compared With Transarterial Chemoembolization in Patients With Large and Unresectable Hepatocellular Carcinoma Staged BCLC A/B
Brief Title: HAIC Versus TACE for Large and Unresectable Hepatocellular Carcinoma Staged BCLC A/B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-170206
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Transarterial Chemoembolization; Large and unresectable HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; Pharmaceutical Preparations; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatic arterial infusion chemotherapy (Experimental): Procedure/Surgery: Hepatic arterial infusion chemotherapy Drug: Folfox Protocol. Hepatic intraarterial infusion via the tumor feeding arteries of Oxaliplatin , fluorouracil, and leucovorin
  Interventions: Procedure: Hepatic arterial infusion; Drug: Folfox Protocol
- Transarterial chemoembolization (Active Comparator): Procedure/Surgery: Transarterial chemoembolization Drug: TACE Drug Protocol. Hepatic intra-arterial infusion with lipiodol mixed with chemotherapy drugs (EADM, lobaplatin, and MMC), and embolization with polyvinyl alcohol particles (PVA)
  Interventions: Procedure: Transarterial chemoembolization; Drug: TACE Drug Protocol

INTERVENTIONS:
Procedure: Hepatic arterial infusion — A standard hepatic artery catheter was introduced via the femoral artery percutaneously. Selective catheterization of the proper hepatic artery was performed using standard diagnostic catheters and fluoroscopic guidance. In the event of multiple arterial supply(including superior-mesenteric artery), the proportion of the liver supplied by each artery was estimated by the arteriogram. After optimal positioning of the catheter in dominant supplying artery to ensure minimal reflux, the catheter was fixed and connected with infusion tube. In the condition of multiple tumors on both left and right lobe, the gastroduodenal artery was embolized and the catheter was positioned in the hepatic proper artery for infusion. Folfox Protocol were infused through the fixed catheter sequentially
  Arms: Hepatic arterial infusion chemotherapy
Procedure: Transarterial chemoembolization — Previous procedure was same with hepatic arterial infusion chemotherapy. After optimal positioning of the catheter, TACE Drug Protocol were injected.
  Arms: Transarterial chemoembolization
Drug: Folfox Protocol — oxaliplatin,leucovorin and 5-FU
  Other Names: Folfox for TAI
  Arms: Hepatic arterial infusion chemotherapy
Drug: TACE Drug Protocol — lipiodol mixed with chemotherapy drugs(EADM , lobaplatin, and MMC) followed by polyvinyl alcohol particles (PVA)
  Other Names: Drugs for transarterial chemotherapy and embolization
  Arms: Transarterial chemoembolization

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) compared with transarterial chemoembolization (TACE) in patients with large and unresectable hepatocellular carcinoma staged BCLC A/B.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients. While a number of studies demonstrate poor effect of TACE for patients with large hepatocellular carcinoma staged BCLC A/B. Our previous prospective study also revealed similar results of large HCC patients treated with TACE. Recently, the results of our preliminary pilot study suggested that, compared with TACE, hepatic arterial infusion chemotherapy (HAIC) may improve tumor response for HCC with large HCC.

Thus, the investigators carried out this prospective nonrandomized control to demonstrate the superiority of HAIC over TACE.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18-75 years;
* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL), simultaneously staged as BCLC A or BCLC B based on Barcelona Clinic Liver Cancer staging system.
* Patients must have at least one tumor lesion that can be accurately measured;
* Solitary tumor with diameter ≥10cm, invaded both left and right lobe; or multiple tumors, diameter of the largest was more than 7cm.
* Diagnosed as unresectable with consensus by the panel of liver surgery experts;
* Re commanded treated by TAI or TACE with consensus by the panel of liver MDT;
* No past history of TACE, TAI, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* No liver protection therapy in 2 weeks before enrolled, and meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin

  ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine

  ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* Poor compliance that can not comply with the course of treatment and follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 16 months
  Best response based on RECIST

SECONDARY OUTCOMES:
Time to progression | 16 months
Adverse Events | 30 Days after HAIC and TACE
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided